CLINICAL TRIAL: NCT03229226
Title: Development and Assessment of a Simulation Model of Focused and Ongoing Professional Practice Evaluations
Acronym: OPPE16
Status: Completed | Type: Observational
Sponsor: Rush University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 15100805-IRB01-AM01
Record Dates: First submitted 2017-07-17; First posted 2017-07-25 (Actual); Last update posted 2017-07-28 (Actual); Status verified 2017-07

CONDITIONS: Competence; Emergencies
Keywords: Simulation; Task Trainer
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 2016 OPPE: All faculty participating in yearly ongoing professional Practice evaluation were eligible for enrollment
  Interventions: Other: Verbal versus procedural assessment

INTERVENTIONS:
Other: Verbal versus procedural assessment — Faculty were assessed on both verbal and simulated performance of procedures.

SUMMARY:
Since 2007, the Joint Commission on Accreditation of Healthcare Organizations (JCAHO) has required evaluation of practicing attending physicians by management to ensure that procedural skills and medical care are meeting the accepted standards of care as assessed by each individual institution. This assessment is known as the ongoing professional practice evaluation (OPPE). There are several methods by which this can be accomplished, including through chart review of clinician practice and by verbally assessing knowledge of the steps required to do a particular procedure. However, for infrequently performed or complicated procedures, these methods may not allow objective evaluation on a regular basis. Simulation using task trainers or manikin models offers an alternative method of objective evaluation in a standardized setting.

The goal of this study is to develop two simulated scenarios to assess physician skill in relatively uncommon procedures and compare the data obtained against the verbal assessment and chart review model previously used at our institution. Two raters will assess each practitioner's verbal and simulated procedures. They will also assess globally their confidence that the physician is capable of performing the procedure safely and correctly based on the verbal or simulated trial.

The investigators anticipate that using a simulated experience for assessment will increase the ability of raters to assess proficiency for the purposes of an OPPE, specifically by increasing the number of critical procedural components that can be objectively evaluated. The investigators hypothesize that there will not be a strong relationship between the scores obtained on the verbal assessment and the scores obtained on the task trainer assessment. The investigators anticipate that there will be a portion of study participants that do not meet a minimum passing standard and may require additional deliberate practice and further testing.

DETAILED DESCRIPTION:
Physician training has developed over recent years to include simulation-based learning as a method of both formative and summative assessment. Simulation based medical education (SBME) with deliberate practice has been shown to be superior to traditional clinical education with respect to procedural skills in physicians in training (McGaghie,W.C. 2011), and a similar concept with Mastery Learning has shown to increase resident skill in lumbar puncture placement. In addition, it has been shown that Simulation Based Mastery Learning (SBML) in central line placement reduces hospital wide rates of central line associated bacterial infections.

When used in continuing medical education (CME), simulation has been shown to be feasible, and to increase clinician confidence in patient management. A recent study of nephrology fellows and attendings in practice showed that both groups scored similarly on a pre-test examination, and that all fellows who completed mastery learning subsequently passed the checklist assessment at the competency level and rated the training session highly.

In other work, simulation has been used for ongoing professional practice assessments (OPPE), for example in psychiatry using online simulated patients and assessments as a way of identifying a smaller number of attendings requiring focused assessment in person). Using electronically collected clinical data, anesthesia cases were reviewed for deviation from the standard of care on several key pieces of documentation common to many anesthesia procedures. This method of direct chart assessment for OPPE may be possible in anesthesia, a field where many cases have similarities in procedure, but would not work for a field such as Emergency Medicine, where the type and acuity of patient encounters varies greatly from day to day.

The ability of Simulation to present a standardized, specific procedural need offers an opportunity to assess Attending Emergency Physicians on a variety of critical procedures in a concise way. The investigators' research aims to present one possible approach to this assessment.

ELIGIBILITY:
Inclusion Criteria:

* Emergency Medicine physician

Exclusion Criteria:

* Not Emergency Medicine physician

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All faculty practicing in an urban emergency department were eligible for enrollment
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2016-05-01 (Actual); Study Completion 2016-05-01 (Actual)

PRIMARY OUTCOMES:
Performance on Procedural Checklist | Immediate
  A 29-item procedural checklist for Central Line and a 21-item procedural checklist for Lumbar puncture will be used to assess performance by clinicians on Central Venous Catheter insertion and Lumbar Puncture performance.

SECONDARY OUTCOMES:
Acceptance of simulated training and assessment format | Immediate
  A survey tool will be used to query participants on their preferred way of both practicing and being assessed on procedural skill. It will also assess whether participants feel inclined to complete a future simulated procedural training session.

CONTACTS AND LOCATIONS:
Overall Officials: Sara M Hock, MD, Principal Investigator — Rush University Medical Center

IPD SHARING:
Plan to Share IPD: Undecided
If requested, data may be shared. Limited generalizability of data may limit its usefulness to other investigators

REFERENCES:
- [Background] OPPE and FPPE: Tools to help make privileging decisions 2013. Wise RA. (Accessed Jul 19, 2017, at http://www.jointcommission.org/jc_physician_blog/oppe_fppe_tools_privileging_decisions/).
- [Background] McGaghie WC, Issenberg SB, Cohen ER, Barsuk JH, Wayne DB. Does simulation-based medical education with deliberate practice yield better results than traditional clinical education? A meta-analytic comparative review of the evidence. Acad Med. 2011 Jun;86(6):706-11. doi: 10.1097/ACM.0b013e318217e119. PMID 21512370
- [Background] Barsuk JH, Cohen ER, Caprio T, McGaghie WC, Simuni T, Wayne DB. Simulation-based education with mastery learning improves residents' lumbar puncture skills. Neurology. 2012 Jul 10;79(2):132-7. doi: 10.1212/WNL.0b013e31825dd39d. Epub 2012 Jun 6. PMID 22675080
- [Background] Barsuk JH, McGaghie WC, Cohen ER, O'Leary KJ, Wayne DB. Simulation-based mastery learning reduces complications during central venous catheter insertion in a medical intensive care unit. Crit Care Med. 2009 Oct;37(10):2697-701. PMID 19885989
- [Background] Barsuk JH, Cohen ER, Potts S, Demo H, Gupta S, Feinglass J, McGaghie WC, Wayne DB. Dissemination of a simulation-based mastery learning intervention reduces central line-associated bloodstream infections. BMJ Qual Saf. 2014 Sep;23(9):749-56. doi: 10.1136/bmjqs-2013-002665. Epub 2014 Mar 14. PMID 24632995
- [Background] Kerr B, Hawkins TL, Herman R, Barnes S, Kaufmann S, Fraser K, Ma IW. Feasibility of scenario-based simulation training versus traditional workshops in continuing medical education: a randomized controlled trial. Med Educ Online. 2013 Jul 18;18:21312. doi: 10.3402/meo.v18i0.21312. PMID 23870304
- [Background] McQuillan RF, Clark E, Zahirieh A, Cohen ER, Paparello JJ, Wayne DB, Barsuk JH. Performance of Temporary Hemodialysis Catheter Insertion by Nephrology Fellows and Attending Nephrologists. Clin J Am Soc Nephrol. 2015 Oct 7;10(10):1767-72. doi: 10.2215/CJN.01720215. Epub 2015 Sep 25. PMID 26408550
- [Background] Barsuk JH, Cohen ER, Nguyen D, Mitra D, O'Hara K, Okuda Y, Feinglass J, Cameron KA, McGaghie WC, Wayne DB. Attending Physician Adherence to a 29-Component Central Venous Catheter Bundle Checklist During Simulated Procedures. Crit Care Med. 2016 Oct;44(10):1871-81. doi: 10.1097/CCM.0000000000001831. PMID 27336437